The Effect of Platelet Rich Plasma on Non-scarring Alopecia

PI: Hooman Khorasani, MD

NCT03689452

**Document Date: 9/21-2018** 

The Effect of Platelet Rich Plasma on Non-scarring Alopecia: A Randomized, Controlled Clinical Trial

PI: Hooman Khorasani, MD

**Date**: 9/21/18

Statistical analyses

Statistical analyses will be performed using SAS version 9.4 (SAS Institute Inc., North Carolina,

United States). Difference scores from baseline to week 8 and from baseline to week 24 will be

calculated for both hair density and caliber. The PRP and saline groups will be compared on

these difference scores using independent samples t-tests. The difference scores will also be

dichotomized based on whether the change over time was positive or negative. The PRP and

saline groups will be compared on these dichotomized scores using chi-square tests. All given p-

values will be two tailed and a p-value of less than 0.05 will be regarded as indicating statistical

significance.